CLINICAL TRIAL: NCT01555502
Title: Health Related Quality of Life After Video Assisted Thoracoscopic Lobectomy for Lung Cancer
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor
Other Study IDs: HRQOL VATS lobectomy
Record Dates: First submitted 2012-03-07; First posted 2012-03-15 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Operable Early Stage NSCLC by the VATS Approach

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- low complications: Patients who had VATS lung resection for NSCLC, and have no or low grade (grade 1 and 2) post operative complications based on the Clavien classification system.
- High complications: Patients who had VATS lung resection for NSCLC, and have no or high grade (grade 3 and 4) post operative complications based on the Clavien classification system.

SUMMARY:
To test the effect of post operative complications on the health related quality of life (HRQOL) after Video Assisted Thoracoscopic Surgery (VATS) for Non-Small Cell Lung Cancer (NSCLC).

The HRQOL of patients with early stage NSCLC will be assessed at baseline (before surgery) using 3 different reliable and valid HRQOL questionnaire (SF-36, EQ-5D and QLQ30/13), then at regular intervals in the early post-operative period (2,4,8 and 12 weeks) the HRQOL will be assessed using the same questionnaires to determine the difference between patients with low/no post operative complications to those with high grade post-operative complications.

Post operative complications will be assess while the patients in the hospital on a daily basis using the Clavien classification system for surgical complications.

ELIGIBILITY:
Inclusion Criteria:

* Adults (more than 18 years)
* early stage NSCLC
* speak English
* No hearing/Speaking difficulties
* Able to walk without assistance
* Surgery via the VATS approach

Exclusion Criteria:

* Less than 18 years old
* Metastatic disease to the lung
* Benign Lung disease
* Advanced NSCLC
* Small Cell Lung Cancer
* Non English speakers
* Walking/Hearing/Speaking difficulties

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with operable early stage NSCLC by the VATS approach who are referred to the Thoracic surgery Center in Edmonton, Alberta, Canada.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Health related Quality of life | Change in health related quality of life at 2 weeks. Change of Health Related Quality of Life at 4 weeks. Change in Health Related Quality of Life at 8 weeks. Change in Health Related Quality of Life at 12 weeks.
  Health Related Quality of Life will be assessed using the SF-36, EQ-5D and QLQ30/13 questionnaires.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Alexandra Hospital, Edmonton, Alberta, Canada